CLINICAL TRIAL: NCT06362031
Title: A Center-Based Chart Review Study to Assess Treatment Outcomes of Venetoclax for the Treatment of Acute Myeloid Leukemia (AML)
Brief Title: A Study to Explore Treatment Patterns, Treatment Outcomes, Healthcare Resource Utilization in Adult Participants With Acute Myeloid Leukemia (AML) Receiving Venetoclax Through Chart Review
Status: Withdrawn | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H18.Oncology.12-SR1812
Record Dates: First submitted 2023-05-31; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Cancer; Venetoclax: Venclyxto; ABT-199
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Venetoclax: Participants with AML receiving venetoclax undergoing chart review.

SUMMARY:
Acute myeloid leukemia (AML), also referred to as acute myelogenous leukemia or acute non-lymphocytic leukemia, is a relatively rare, yet aggressive, type of cancer. This study will evaluate treatment patterns, treatment outcomes, healthcare resource utilization in adult participants with AML receiving venetoclax.

Data from up to 700 participants will be collected. No participants will be enrolled in this study.

Participants' charts will be reviewed. No drug will be administered as a part of this study. The duration of the observation period is up to 10 months.

There is no additional burden for participants in this trial. All visits must be completed prior to data extraction and participants will be followed for up to 10 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant received a diagnosis for acute myeloid leukemia (AML).
* The participant was initiated on the studied line of therapy for previously untreated AML, as noted in the protocol.
* The participant was treated with the studied line of therapy at least 28 days prior to date of data collection.
* Information on the participant's treatments, selected (or important) clinical characteristics, and outcomes is available from the start of the studied line of therapy onwards.

Exclusion Criteria:

* The participant received the studied line of therapy as part of a clinical trial.
* Participant received prior lines of therapy for AML.
* The participant has a history of malignancies within 2 years prior to the studied line of therapy, other than AML, and with the exception of what is noted in the protocol.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Participants with Acute Myeloid Leukemia (AML) being treated with venetoclax.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 10 Months
  OS will be measured as the number of days between the initiation of the studied line of therapy and death.
Event-free survival (EFS) | Up to 10 Months
  EFS will be measured as the number of days between the initiation of the studied line of therapy and disease progression, or refractory disease, or death.
Percentage of Participants Achieving Best Overall Response | Up to 10 Months
  Physician-reported best response achieved from initiation of the studied line of therapy until the earliest of disease progression, refractory disease, relapse, switch to a new line of therapy, or end of follow-up or death.
Duration of Response (DoR) | Up to 10 Months
  DoR is is defined as complete remission (CR), complete remission with incomplete marrow recovery (CRi), complete remission with partial hematologic recovery (CRh), morphologic leukemia-free state (MLFS); in days.
Percentage of Participants with Transfusion Independence (TI) | Up to 10 Months
  TI from initiation of the studied line of therapy until disease progression, refractory disease, relapse, or switch to a new line of therapy.

SECONDARY OUTCOMES:
Number of Participants with Healthcare Resource Utilization (HRU) | Up to 10 Months
  HRU is measured from initiation of the studied line of therapy until physician recorded disease progression, refractory disease, relapse, or switch to a new line of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H18.Oncology.12-SR1812